CLINICAL TRIAL: NCT02373020
Title: ROLE OF E COLI IN Colorectal Tumourigenesis
Brief Title: Enteropathogenic Escherichia Coli (EPEC): Does it Have a Role in Colorectal Tumourigenesis?
Acronym: EPEC
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, MOHAMED ABDELLATIF, consultant, Mansoura University
Other Study IDs: e coli
Record Dates: First submitted 2015-02-16; First posted 2015-02-26 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-02

CONDITIONS: Enteropathogenic Escherichia Coli .; Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months

GROUPS / COHORTS (2):
- group 1: colonoscopic biopsies from patients with colorectal cancer patients
  Interventions: Other: colonoscopic biopsies
- (Group 2: colonoscopic biopsies from healthy controls
  Interventions: Other: colonoscopic biopsies

INTERVENTIONS:
Other: colonoscopic biopsies

SUMMARY:
Despite the characterization of many aetiologic genetic changes. The specific causative factors in the development of sporadic colorectal cancer remain unclear. This study was performed to detect the possible role of Enteropathogenic Escherichia coli (EPEC) in developing colorectal carcinoma.

DETAILED DESCRIPTION:
Fresh biopsy specimens have been obtained from the colonic mucosa overlying the colorectal cancer as well as from the colon of the healthy controls. Culture, genotyping and virulence of EPEC were done using (nutrient broth culture, and PCR). Strains biochemically identified as E. coli were selected from the surface of a MacConkey's plate and were serogrouped by slide agglutination tests

ELIGIBILITY:
Inclusion Criteria:

* patients with colorectal carcinoma after have been diagnosed

Exclusion Criteria:

* Patients with inflammatory bowel disease (IBD) or macroscopic signs of inflammation were excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients who were diagnosed to have colorectal cancer (Group 1) and healthy controls who had colonoscopy for colorectal symptoms in the same study period (Group 2
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
virulence genes: eaeA, bfpA and stx. PCR | 1 week
  E. coli colonies isolated from the mucosa of colorectal cancers and from healthy controls were harvested and subjected to DNA extraction (QIAGEN)

SECONDARY OUTCOMES:
EPEC serogrouping: | 1 week
  Strains biochemically identified as E. coli were selected from the surface of a MacConkey's plate and were serogrouped by slide agglutination tests to detect EPEC using O-specific nonavalent E.coli antiserum (O26, O55, O86, O111, O114, O119, O124, O125, O126, O127, O128, O142), according to the manufacturer's instructions (Bio-Rad).
Strains: OF E COLI | 1 week
  The specimens were immediately transferred to the lab, inoculated in nutrient broth and vortexed for a few seconds then incubated overnight. The following day the broth culture was subcultured on enteric isolation media. Identification of E. coli was carried out by using standard biochemical methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt